CLINICAL TRIAL: NCT03310385
Title: Efficacy and Safety of GHX02 in the Treatment of Acute Bronchitis: a Phase 2, Double-blind, Randomized Placebo-controlled Trial
Brief Title: Efficacy and Safety of GHX02 in the Treatment of Acute Bronchitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daejeon University (Other)
Responsible Party: Principal Investigator, Yang Chun Park, Professor, Daejeon University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DJRM-2017-01
Record Dates: First submitted 2017-10-06; First posted 2017-10-16 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Acute Bronchitis
Keywords: Acute Bronchitis, Herbal Medicine
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Intervention Model Description: multicentre, dose-finding,double-blind, randomized placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose GHX02 group(1,920mg/day) (Experimental): 4 tablets of the GHX02, three times daily for 7 days
  Interventions: Drug: GHX02
- Standard-dose GHX02 group(960mg/day) (Experimental): 2 tablets of the GHX02 and 2 tablets of the placebo, three times daily for 7 days
  Interventions: Drug: GHX02; Drug: Placebo
- Placebo control (Placebo Comparator): 4 tablets of the placebo, three times daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GHX02 — Herbal medicine originating from gualouhengryunhwan
  Arms: High-dose GHX02 group(1,920mg/day); Standard-dose GHX02 group(960mg/day)
Drug: Placebo — Placebo tablets
  Arms: Placebo control; Standard-dose GHX02 group(960mg/day)

SUMMARY:
This study is a phase 2, multicentre, dose-finding, double-blind, randomized placebo-controlled trial to evaluate the efficacy and safety of two different doses of GHX02, compared with placebo, for acute bronchitis. One-hundred and fifty patients will be included in this trial and randomly assigned to either a high-dose GHX02 group(1920mg/day), standard-dose GHX02 group(960mg/day), or control group(placebo) in a 1:1:1 allocation ratio. Patients will take one of the medications three times a day for 7 days, with 3 visiting days(screening, day0, day7). On the screening day, the Korean Standard Tool of Pattern Identification of Cough and Sputum, a diagnostic system that determines therapy in Traditional Korean Medicine, will be used to allocate patients into three groups of wind-heat, wind-cold or others.

ELIGIBILITY:
Inclusion Criteria:

1. age 19-75 years
2. BSS ≥ 5 points at visit2 due to acute bronchitis
3. symptoms starting within 2 weeks before study inclusion
4. patients who consent to participate

Exclusion Criteria:

1. pregnant or breast-feeding
2. treatment with antibiotics, bronchodilators, glucocorticoids, immune-depressants, or other clinical trial medicines during the last 4 weeks before study inclusion
3. treatment with antitussives or expectorants during the last 7 days before study inclusion
4. history or presence of confounding respiratory disease that may affect evaluation of the efficacy of clinical medicine (e.g. chronic bronchitis, chronic obstructive pulmonary disease (COPD), bronchiectasis, asthma, pneumonia, cystic fibrosis, lung cancer, or active pulmonary tuberculosis)
5. liver or renal impairment (alanine aminotransferase(ALT), aspartate aminotransferase(AST), alkaline phosphatase(ALP) ≥ 3 times the normal upper limit, or creatinine> 3.0 mg/dL at screening)
6. history or presence of clinically relevant cardiovascular, renal, metabolic, haematological, neurological, psychiatric, systemic, infectious disease, or malignant tumour(except where there is no recurrence for more than 5 years after surgery)
7. history of alcoholism or substance abuse
8. participation in other clinical drug(medicine) trials during the last 30 days before study inclusion
9. judged by the investigators to be inappropriate for the clinical trial.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-03-18 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in BSS(Bronchitis Severity Score) | Day0, Day7
  BSS comprises the sum of five major symptom scores for acute bronchitis: cough, sputum, dyspnea, chest pain during coughing, and rales on auscultation. Each symptom is scored on a 4-point-scale (0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe), with a maximum total score of 20 points. The investigator assesses symptom scores on the basis of the patient's subjective symptoms.

SECONDARY OUTCOMES:
Change in Questionnaire of Clinical Symptoms of Cough and Sputum | Day0, Day7
  Questionnaire items are as follows: (1) cough -frequency, intensity, sensitivity; (2) sputum -frequency, volume, difficulty to cough-up, appearance, color; (3) activities of daily living; (4) night-time sleeping. Each item is scored on a 4-point-scale, with a total maximum score of 40 points.
Change in Leicester Cough Questionnaire-acute(LCQ-acute) | Day0, Day7
  It consists of 19 items divided into three parts, physical, psychological, and social, each scored from 1 to 7. The total score is the sum of the average scores(1-7 points) for each part. The higher the score, the better the quality of life.
Change in frequency of coughing fits | Day0, Day1, Day2, Day3, Day4, Day5, Day6, Day7
  participants will be classified into one of the following scales: 0 = 0 time/day, 1 = 1 time/day, 2 = 2-3 times/day, 3 = 4-5 times/day(sometimes), 4 = 6-10 times/day(frequent), 5 = over 15 times/day(consistently).
Integrative Medicine Outcome Scale(IMOS) | Day7
  It's a 5-point-scale for evaluating improvement after treatment (where, 1=complete recovery, 2=major improvement, 3=slight-to-moderate improvement, 4=no change, 5=deterioration), either by the patient or investigator (the investigator in this trial).
Integrative Medicine Patient Satisfaction Scale(IMPSS) | Day7
  It's a 5-point-scale for evaluating patient satisfaction with the treatment (where, 1=very satisfied, 2=satisfied, 3=neutral, 4=dissatisfied, 5=very dissatisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Dunsan Korean Medicine Hospital, Daejeon University, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Ji KY, Kim KM, Oh JJ, Kim JW, Lee WJ, Cho H, Lee HK, Lee JY, Chae S. Assessment of the 4-week repeated-dose oral toxicity and genotoxicity of GHX02. J Appl Toxicol. 2020 Feb;40(2):270-284. doi: 10.1002/jat.3902. Epub 2019 Sep 12. PMID 31515828
- [Derived] Lyu YR, Yang WK, Park SJ, Kim SH, Kang WC, Jung IC, Park YC. Efficacy and safety of GHX02 in the treatment of acute bronchitis: protocol of a phase II, double-blind, randomised placebo-controlled trial. BMJ Open. 2018 May 14;8(5):e019897. doi: 10.1136/bmjopen-2017-019897. PMID 29764875